CLINICAL TRIAL: NCT02499991
Title: Memory Intervention for Older Adults - A Pilot Study
Brief Title: Memory Intervention for Older Adults - (Social)
Acronym: Social
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Daniel Saltel, Community Health Science Msc Student, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2015:243
Record Dates: First submitted 2015-07-10; First posted 2015-07-16 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Memory Impairment
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Treatment group will keep diary of social events according to training instructions.
  Memory intervention will be used.
  Interventions: Behavioral: memory
- Control (No Intervention): Control group will use own memory of social events without training instructions.

INTERVENTIONS:
Behavioral: memory — keep track of social events in diary for memory recall. Used by treatment group
  Arms: Treatment

SUMMARY:
Research shows that there are a plenitude of interventions that can be used to enhance memory for older adults; however, the evidence as to whether these interventions enhance memory for daily activities is equivocal. The purpose of this pilot study is to test a memory intervention that is potentially useful in everyday life. Objectives of the pilot study are: 1) to examine the feasibility of the intervention (e.g., ease of use of materials provided); and 2) to gain preliminary evidence of the intervention's impact on recall of recent daily social events. Participants will be 20 cognitively healthy (i.e. not cognitively impaired) older adults, with 10 participants randomly assigned to either an intervention or control group, respectively. The study will consist of: a) a pre-training session; b) seven days of independent memory training; and c) a post-training session. The pre-training session will involve a test that measures recall of daily social events from the previous week. This will be followed by seven days of training for recall of daily social events. During the seven days, the intervention group will perform daily memory tasks using self-instructional materials given to them by the researcher, whereas the control group will use their own strategies for remembering social events that they are involved in during the week. The post-training session will occur after the seven days and will involve the same test as the pre-training session that measures recall of social events from the previous week. The hypotheses are that: a) recall of social events will be higher for the post-training test than in the pre-training test and; b) recall will be better for in the intervention group than the control group. The ease of use of the memory recall materials provided to the intervention group will be assessed in interviews.

DETAILED DESCRIPTION:
Method Participants The sample will consist of 20 cognitively healthy older adults (aged 55 or older) recruited from the Centre on Aging participant database. The participant database has been approved by the Health REB (REB #HS14652). Individuals who are in the participant database have given their consent to be contacted by researchers about their willingness to participate in specific research projects. Names of individuals are provided to researchers by the Centre on Aging upon submission of REB approval and the research protocol.

Materials Questionnaires Pre-training Questionnaire - demographics. The questionnaire will consist of general questions about the participants. Items will include gender, age, and experience with memory training.

Pre-training memory recall test. The questionnaire will ask participants to describe social events they did during the previous week. This questionnaire will be given in the pre-training session.

Post-training memory recall test. The questionnaire will ask participants to describe social events they did during the previous week. This questionnaire will be given in the post-training session.

Post-training questionnaire. The questionnaire will ask participants about their thoughts regarding the format and usefulness of the instruction materials. For example, participants will be asked if they thought the study helped them remember social events.

Intervention group materials Memory tasks - instructions. This document instructs participants in the intervention group on how to use the memory tasks for daily social events.

Memory tasks - forms. Each day has a separate document that has a) a diary of social events; and b) tasks to review the week's social events.

Memory tasks - forms example. This is an example of the above form filled out to help explain how memory tasks are to be done.

Design This study involves an experimental design, whereby participants will be randomly assigned to one of two groups, an intervention group (n=10) and a control group (n=10). The independent variable is, therefore, the presence or absence of the daily memory recording task for social events. The dependent variables are: (a) the changes in performance on the written recall tests from pre- to post-training; and (b) the difference between the groups (i.e., Control vs. intervention group) on performance of memory of social events. Information about how useful the intervention materials were will be used in a more qualitative way to help improve the intervention.

Procedure The study will consist of: a) a pre-training session; b) seven days of independent memory training (intervention group) or usual way of remembering social events (control group); and c) a post-training session. The pre-training session will involve a test that measures recall of social events from the previous week. This will be followed by seven days of training for recall of daily social events. The post-training session will occur after the seven days and involve the same test as the pre-training session that measures recall of social events from the previous week.

Pre-training session. There will be separate pre-training sessions for each individual participant with the principal investigator either at the University of Manitoba (Bannatyne campus or Fort Garry campus) or, if participants prefers, in his or her own home. During the pre-training session, the principal investigator will provide an informed consent form to the participant. The principal investigator will describe the project, review the consent form and answer any questions. Once the participant provides written consent, a demographics questionnaire will be administered. A pre-training memory recall test will also be done that asks participants to list social events they did during the previous week.

Seven day training week. Materials will be provided to the intervention group during the pre-training session. Materials will include: a) instructions for memory tasks; b) forms for each day for diaries and tasks; and c) an example of the form filled out. The control group will not receive materials and will have to rely on their own memory strategies to remember social events during the 7 days.

Post-training session. There will be separate post-training sessions for each individual participant with the principal investigator either at the University of Manitoba (Bannatyne campus or Fort Garry campus) or in the participants' homes. A post-training memory recall test will be done that asks participants to list social events that they did on the previous week (i.e., this is the same test that was used in pre-training session). The post-training questionnaire will then also be administered to each participants.

Data Management Data will be entered into the computer. The computer file will not contain any names or addresses and each participant data will be identified by a unique participant ID only. Consent forms will be stored in a locked filing cabinet in Dr. Menec's research space (S112 Medical Services Bldg).

Analyses A total score of all social events recalled will be created. Scores will be calculated by the following scheme: a) one point for remembering an event; and b) one point for remembering the day of the event. Other scoring approaches will also be considered; for example, assigning a higher score if more detail about a person met is remembered. SPSS will be used to test hypotheses using two independent group t-tests. The use of t-tests is justified because a) the investigators can compare scoring on pre- and post-session memory recall tests; b) the investigators have an appropriate sample size of 20; and c) the investigators have two independent groups. The usefulness of the memory intervention materials will be examined more qualitatively by looking at responses to each of the questions and participants' comments.

ELIGIBILITY:
Inclusion Criteria:

* cognitively healthy

Exclusion Criteria:

* diagnosed cognition impairments such as Alzheimer's

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Memory Recall Test (change from first session to second session i.e., 7 days later) | First session, second session (7 days later from first session)
  The questionnaire will ask participants to describe social events they did during the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: Verena Menec, Phd, Study Director — University of Manitoba